CLINICAL TRIAL: NCT03496948
Title: PAD-TeGeCoach: Health Coaching and Telemetry Supported Walking Exercise for Improving Quality of Life
Brief Title: Telephone Health Coaching and Remote Exercise Monitoring for Peripheral Artery Disease
Acronym: TeGeCoach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tegecoach; 01NVF17013 (Other Grant/Funding Number: German Innovation Fund (Innovationsfonds))
Record Dates: First submitted 2018-03-23; First posted 2018-04-12 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Peripheral Artery Disease; Atherosclerosis; Peripheral Arterial Disease; Arterial Occlusive Diseases; Vascular Diseases; Peripheral Vascular Diseases; Cardiovascular Diseases
Keywords: PAD; Peripheral Artery Disease; Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Peripheral Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Study arms: TeGeCoach (Intervention); Treatment-as-Usual (TAU)
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TeGeCoach (Experimental): Home-based exercise program consisting of telephone health coaching, remote walking exercise monitoring based on wearable monitors and intensified primary care.
  Interventions: Behavioral: TeGeCoach
- Usual care group (TAU) (No Intervention): Patients randomized to TAU receive written information about courses offered by their statutory health insurance. Health insurance companies offer a variety of courses to encourage regular exercise and to promote lifestyle changes, including SEPs (vascular and cardio exercise), physical therapy, nutritional assistance programs, smoking cessation programs, weight loss programs, and patient education programs for obesity and diabetes.

INTERVENTIONS:
Behavioral: TeGeCoach — 12-month long telephone health coaching carried out by specially trained coaches. The health coaching is a patient-centered approach based on motivational interviewing, shared decision-making and active listening techniques. Primary care physicians will be constantly involved receiving regular health reports from the coach.
  The walking exercise is based on the principle of interval training. Patients will continuously wear an activity monitor device to review their exercise performance and for remote exercise monitoring by the coach. This activity information will be regularly reviewed by the coach to ensure that the patient adheres to the individual walking exercise prescription.
  Arms: TeGeCoach

SUMMARY:
Peripheral artery disease (PAD) is the third most prevalent cardiovascular disease worldwide, with over 200 million people affected. Most prominent symptom is leg pain while walking known as intermittent claudication. Based on the currently existing gaps in the management of intermittent claudication, the objective of the this study is to explore the clinical effectiveness and cost advantage of TeGeCoach, a 12-month long home-based exercise program, compared to usual care. TeGeCoach consists of telephone health coaching, remote walking exercise monitoring based on wearable activity monitors and intensified primary care. It is hypothesized that TeGeCoach will improve functional outcomes and will reduce total health care costs.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is the third most prevalent cardiovascular disease worldwide and has become a serious public health issue, with over 200 million people affected. Smoking and diabetes are the strongest risk factors for the development of peripheral artery disease, but also high cholesterol, high blood pressure and sedentary lifestyle. The most prominent symptom is leg pain while walking known as intermittent claudication, as the muscles do not get enough blood during exercise to meet the needs. To improve mobility, first line treatment for intermittent claudication are outpatient supervised exercise programs (SEPs); however, their implementation face manifold challenges: low patient adherence, no reimbursement by insurers, high costs of course implementation, and low course availability. These barriers led to the development of home-based exercise programs, which are similarly effective when combined with a structured approach by setting exercise goals, monitoring exercise activity, and regular follow up with a coach. Therefore, this trial aims to determine the clinical effectiveness and cost advantage of TeGeCoach, a 12-month long structured home-based exercise program (HEP), compared with usual care of intermittent claudication. It is hypothesized that TeGeCoach will improve walking impairment and will lower the need of health care resources that are spent on patients with PAD at 24-month follow-up.

The investigators will conduct a prospective, open-label, pragmatic randomized controlled clinical trial in a health insurance setting. 1760 patients with peripheral artery disease at Fontaine stage II will be randomly assigned either to TeGeCoach or Care-as-usual (usual care). TeGeCoach consists of telemonitored walking exercise using wearable activity trackers, telephone health coaching and medical supervision by a physician. The health coaching is a patient-centered approach based on motivational interviewing, shared decision-making and active listening techniques for supporting better patient engagement and activation, disease self-care, treatment adherence and lifestyle management. Depending on the individual functional status and exercise capacity, participants will be asked to walk up to seven times a week. Usual care participants regularly receive information leaflets and can access supervised exercise programs, physical therapy and a variety of programs for promoting a healthy lifestyle. Primary outcomes are functional capacity measured by the Walking Impairment Questionnaire (WIQ). Secondary outcome measures include quality of life, health literacy and health behavior. Claims data is used to collect total health care costs, healthcare resource use and (severe) adverse events. Outcomes will be measured at three time points (0, 12, and 24 months).

Clearly, the current routine care of intermittent claudication in patients with PAD is partly ineffective und insufficient, with the consequence of a poorly served patient population and worsening disease condition. TeGeCoach may provide an effective and feasible alternative in the management of intermittent claudication by improving access to supervised exercise while at the same time potentially reducing health care costs.

ELIGIBILITY:
Inclusion Criteria:

* Insured with one of the three participating health insurance companies
* Sufficient German language skills to follow the telephone-based health coaching
* Access to a telephone (landline or mobile);
* Primary or secondary diagnosis of PAD at Fontaine stage IIa or IIb within the last 36 months, but no primary or secondary diagnosis of PAD at Fontaine stage I within the last 12 months; or at Fontaine stage III or IV within the last 36 months

Inpatient and outpatient diagnoses from routine statutory health insurance data will be used to identify eligible patients.

Exclusion Criteria:

* Immobility that goes beyond claudication (inability to carry out intervention and competing risks)
* Severe and persistent mental disorders (adherence reasons)
* Suicidality (safety reasons)
* Life-threatening somatic diseases (e.g., cancer; competing risk)
* Active or recent participation in any other PAD intervention trial
* Ongoing hospitalization; alcoholism and other drug dependency (adherence reasons)
* Heart failure graded New York Heart Association (NYHA) class III and IV (inability to carry out intervention and competing risks)

Ineligible patients are identified based on diagnoses that were made in inpatient settings only, given the considerable number of diagnostic errors in outpatient settings.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1982 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Change in score on Walking Impairment Questionnaire (WIQ) | baseline, 12-month and 24-month follow-up
  The patient-reported WIQ is a valid clinical tool to classify patient-perceived walking impairment in patients with PAD in terms of pain, walking speed, walking distance and the climbing of stairs. The WIQ has been shown to be responsive to treatment effects and thus can be used as an alternative to treadmill testing for an objective assessment of walking claudication.

SECONDARY OUTCOMES:
Change in score on Walking Estimated Limitation Calculated by History (WELCH) questionnaire | baseline, 12-month and 24-month follow-up
  The WELCH is a four-item questionnaire to estimate walking limitation in patients with suspected peripheral artery disease.
Change in score on EQ5D-5L questionnaire | baseline, 12-month and 24-month follow-up
  The EQ5D-5L is a standardized instrument developed by the EuroQoL Group for the measurement of health-related quality of life. There are five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ5D-5L has been validated for the general German population.
Change in score on Short Form Health Survey (SF-12) | baseline, 12-month and 24-month follow-up
  The SF-12 is a self-report questionnaire for the measurement of generic health status involving multiple health dimensions: physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems and mental health. SF-12 is a short version of the SF-36, with good psychometric properties. The German version has been cross-validated with the original English version.
Change in score on Vascular Quality of Life Questionnaire (VascuQoL-25) | baseline, 12-month and 24-month follow-up
  The VascuQol-25 is a highly-responsive validated questionnaire for the measurement of PAD-specific health-related quality of life, with a high level of construct and convergence validity. The questionnaire consists of five domains (Activity, Symptom, Pain, Emotional and Social) and has 25 items in total.
Change in score on Patient Health Questionnaire (PHQ-9) | baseline, 12-month and 24-month follow-up
  The PHQ-9 is a brief valid questionnaire for the diagnosis of depression that can also be used to identify depression outcome measures and changes over time. The German version has been validated twice.
Change in score on Generalized Anxiety Disorder (GAD-7) questionnaire | baseline, 12-month and 24-month follow-up
  The GAD-7 is brief questionnaire for the detection of Generalized Anxiety Disorder, which has been validated in primary care setting and in the general population.
Change in score on Alcohol Use Disorders Identification Test (AUDIT-C) | baseline, 12-month and 24-month follow-up
  The AUDIT-C is a brief screening instrument to identify harmful alcohol consumption, consisting of three questions. Regarding its psychometric properties, the AUDIT-C has been shown to be reliable and valid instrument to screen alcohol misuse in primary care settings.
Change in score on Fagerström Test for Nicotine Dependence (FTND) | baseline, 12-month and 24-month follow-up
  To identify tobacco dependence, the 6-item long Fagerström Test for Nicotine Dependence (FTND) will be used, which has been shown to be validly assessing the physical addiction to nicotine.
Change in score on Health Literacy Questionnaire (HLQ) | baseline, 12-month and 24-month follow-up
  The HLQ is a comprehensive tool with excellent psychometric properties for the measurement of health literacy. The HLQ examines nine dimensions of health literacy.
Change in score on Patient Activation Measure (PAM-13) | baseline, 12-month and 24-month follow-up
  PAM-13 has been shown to be a valuable tool for the measurement of patient activation by dividing people into one of four activation levels. The German version has been validated, with good psychometric properties.
Change in utilization of medical services | baseline, 12-month and 24-month follow-up
  Routine health insurance data: time period until hospitalization; probability of hospitalization; number and duration of inpatient hospitalization; outpatient medical treatment; drug dose (defined daily dose - DDD).
Change in severe (adverse) events | baseline, 12-month and 24-month follow-up
  Routine health insurance data: death, amputation, revascularization, etc.
Change in total health care costs | baseline, 12-month and 24-month follow-up
  Routine health insurance data: hospital billing and insurance reimbursement; inpatient hospital cost; inpatient rehabilitation costs; ambulatory care costs; costs for drugs and other medical supplies; sick pay costs.

OTHER OUTCOMES:
Questionnaire on Satisfaction in Outpatient Care (ZAPA; intervention arm only) | 12-month follow-up
  ZAPA is a brief (4 items) and psychometrically valid German questionnaire for measuring the patient's global satisfaction with his or her outpatient care, including the quality and extent of information received and his/her involvement in clinical decisions (i.e. shared-decision making).
Change in exercise adherence (intervention arm only) | baseline and 12-month follow-up
  Activity tracker data: e.g. number of alerts and corresponding phone calls made when step frequency or the duration of exercise sessions fall below an individual threshold range, amount of steps, net walking time (> 50 steps/minute) per day/week
Change in amount of steps/net walking time (intervention arm only) | baseline and 12-month follow-up
  Coaching software data

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Dirmaier, PD Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Frank Bienert, Study Director — KKH statutory health insurance; Lutz Herbarth, Dr., Study Chair — KKH statutory health insurance
Locations (3):
- Germany (3):
  - TK statutory health insurance, Hamburg
  - KKH statutory health insurance, Hanover
  - Mhplus Statutory Health Insurance, Nuremberg

IPD SHARING:
Plan to Share IPD: Yes
It is planned to share all individual participant data (IPD) that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: After study completion
Access Criteria: Available upon request

REFERENCES:
- [Background] Fowkes FG, Rudan D, Rudan I, Aboyans V, Denenberg JO, McDermott MM, Norman PE, Sampson UK, Williams LJ, Mensah GA, Criqui MH. Comparison of global estimates of prevalence and risk factors for peripheral artery disease in 2000 and 2010: a systematic review and analysis. Lancet. 2013 Oct 19;382(9901):1329-40. doi: 10.1016/S0140-6736(13)61249-0. Epub 2013 Aug 1. PMID 23915883
- [Background] Criqui MH, Aboyans V. Epidemiology of peripheral artery disease. Circ Res. 2015 Apr 24;116(9):1509-26. doi: 10.1161/CIRCRESAHA.116.303849. PMID 25908725
- [Background] Sampson UK, Fowkes FG, McDermott MM, Criqui MH, Aboyans V, Norman PE, Forouzanfar MH, Naghavi M, Song Y, Harrell FE Jr, Denenberg JO, Mensah GA, Ezzati M, Murray C. Global and regional burden of death and disability from peripheral artery disease: 21 world regions, 1990 to 2010. Glob Heart. 2014 Mar;9(1):145-158.e21. doi: 10.1016/j.gheart.2013.12.008. PMID 25432124
- [Background] Gerhard-Herman MD, Gornik HL, Barrett C, Barshes NR, Corriere MA, Drachman DE, Fleisher LA, Fowkes FG, Hamburg NM, Kinlay S, Lookstein R, Misra S, Mureebe L, Olin JW, Patel RA, Regensteiner JG, Schanzer A, Shishehbor MH, Stewart KJ, Treat-Jacobson D, Walsh ME. 2016 AHA/ACC Guideline on the Management of Patients With Lower Extremity Peripheral Artery Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2017 Mar 21;135(12):e726-e779. doi: 10.1161/CIR.0000000000000471. Epub 2016 Nov 13. PMID 27840333
- [Background] Berger JS, Ladapo JA. Underuse of Prevention and Lifestyle Counseling in Patients With Peripheral Artery Disease. J Am Coll Cardiol. 2017 May 9;69(18):2293-2300. doi: 10.1016/j.jacc.2017.02.064. PMID 28473134
- [Background] Makris GC, Lattimer CR, Lavida A, Geroulakos G. Availability of supervised exercise programs and the role of structured home-based exercise in peripheral arterial disease. Eur J Vasc Endovasc Surg. 2012 Dec;44(6):569-75; discussion 576. doi: 10.1016/j.ejvs.2012.09.009. Epub 2012 Sep 30. PMID 23034408
- [Background] Harwood AE, Smith GE, Cayton T, Broadbent E, Chetter IC. A Systematic Review of the Uptake and Adherence Rates to Supervised Exercise Programs in Patients with Intermittent Claudication. Ann Vasc Surg. 2016 Jul;34:280-9. doi: 10.1016/j.avsg.2016.02.009. Epub 2016 Apr 25. PMID 27126713
- [Background] McDermott MM, Polonsky TS. Home-Based Exercise: A Therapeutic Option for Peripheral Artery Disease. Circulation. 2016 Oct 18;134(16):1127-1129. doi: 10.1161/CIRCULATIONAHA.116.023691. No abstract available. PMID 27754945
- [Background] Collins TC, Lunos S, Carlson T, Henderson K, Lightbourne M, Nelson B, Hodges JS. Effects of a home-based walking intervention on mobility and quality of life in people with diabetes and peripheral arterial disease: a randomized controlled trial. Diabetes Care. 2011 Oct;34(10):2174-9. doi: 10.2337/dc10-2399. Epub 2011 Aug 26. PMID 21873560
- [Background] Fakhry F, Spronk S, de Ridder M, den Hoed PT, Hunink MG. Long-term effects of structured home-based exercise program on functional capacity and quality of life in patients with intermittent claudication. Arch Phys Med Rehabil. 2011 Jul;92(7):1066-73. doi: 10.1016/j.apmr.2011.02.007. PMID 21704786
- [Background] Gardner AW, Parker DE, Montgomery PS, Blevins SM. Step-monitored home exercise improves ambulation, vascular function, and inflammation in symptomatic patients with peripheral artery disease: a randomized controlled trial. J Am Heart Assoc. 2014 Sep 18;3(5):e001107. doi: 10.1161/JAHA.114.001107. PMID 25237048
- [Background] Gardner AW, Parker DE, Montgomery PS, Scott KJ, Blevins SM. Efficacy of quantified home-based exercise and supervised exercise in patients with intermittent claudication: a randomized controlled trial. Circulation. 2011 Feb 8;123(5):491-8. doi: 10.1161/CIRCULATIONAHA.110.963066. Epub 2011 Jan 24. PMID 21262997
- [Background] Parmenter BJ, Dieberg G, Smart NA. Exercise training for management of peripheral arterial disease: a systematic review and meta-analysis. Sports Med. 2015 Feb;45(2):231-44. doi: 10.1007/s40279-014-0261-z. PMID 25230780
- [Background] Al-Jundi W, Madbak K, Beard JD, Nawaz S, Tew GA. Systematic review of home-based exercise programmes for individuals with intermittent claudication. Eur J Vasc Endovasc Surg. 2013 Dec;46(6):690-706. doi: 10.1016/j.ejvs.2013.09.004. Epub 2013 Sep 11. PMID 24076079
- [Background] Fokkenrood HJ, Bendermacher BL, Lauret GJ, Willigendael EM, Prins MH, Teijink JA. Supervised exercise therapy versus non-supervised exercise therapy for intermittent claudication. Cochrane Database Syst Rev. 2013 Aug 23;(8):CD005263. doi: 10.1002/14651858.CD005263.pub3. PMID 23970372
- [Background] Normahani P, Kwasnicki R, Bicknell C, Allen L, Jenkins MP, Gibbs R, Cheshire N, Darzi A, Riga C. Wearable Sensor Technology Efficacy in Peripheral Vascular Disease (wSTEP): A Randomized Controlled Trial. Ann Surg. 2018 Dec;268(6):1113-1118. doi: 10.1097/SLA.0000000000002300. PMID 28498233
- [Background] McDermott MM, Domanchuk K, Liu K, Guralnik JM, Tian L, Criqui MH, Ferrucci L, Kibbe M, Jones DL, Pearce WH, Zhao L, Spring B, Rejeski WJ. The Group Oriented Arterial Leg Study (GOALS) to improve walking performance in patients with peripheral arterial disease. Contemp Clin Trials. 2012 Nov;33(6):1311-20. doi: 10.1016/j.cct.2012.08.001. Epub 2012 Aug 7. PMID 23158112
- [Background] McDermott MM, Guralnik JM, Criqui MH, Ferrucci L, Zhao L, Liu K, Domanchuk K, Spring B, Tian L, Kibbe M, Liao Y, Lloyd Jones D, Rejeski WJ. Home-based walking exercise in peripheral artery disease: 12-month follow-up of the GOALS randomized trial. J Am Heart Assoc. 2014 May 21;3(3):e000711. doi: 10.1161/JAHA.113.000711. PMID 24850615
- [Background] Harter M, Dirmaier J, Dwinger S, Kriston L, Herbarth L, Siegmund-Schultze E, Bermejo I, Matschinger H, Heider D, Konig HH. Effectiveness of Telephone-Based Health Coaching for Patients with Chronic Conditions: A Randomised Controlled Trial. PLoS One. 2016 Sep 15;11(9):e0161269. doi: 10.1371/journal.pone.0161269. eCollection 2016. PMID 27632360
- [Background] Kivela K, Elo S, Kyngas H, Kaariainen M. The effects of health coaching on adult patients with chronic diseases: a systematic review. Patient Educ Couns. 2014 Nov;97(2):147-57. doi: 10.1016/j.pec.2014.07.026. Epub 2014 Aug 1. PMID 25127667
- [Background] Rejeski WJ, Spring B, Domanchuk K, Tao H, Tian L, Zhao L, McDermott MM. A group-mediated, home-based physical activity intervention for patients with peripheral artery disease: effects on social and psychological function. J Transl Med. 2014 Jan 28;12:29. doi: 10.1186/1479-5876-12-29. PMID 24467875
- [Derived] Heider D, Rezvani F, Matschinger H, Dirmaier J, Harter M, Herbarth L, Steinisch P, Bobinger H, Schuhmann F, Krack G, Korth T, Thomsen L, Chase DP, Schreiber R, Alscher MD, Finger B, Konig HH. The effect of telephone health coaching and remote exercise monitoring for peripheral artery disease (TeGeCoach) on health care cost and utilization: results of a randomized controlled trial. Eur J Health Econ. 2024 Jun;25(4):615-629. doi: 10.1007/s10198-023-01616-4. Epub 2023 Jul 10. PMID 37428355
- [Derived] Rezvani F, Heider D, Harter M, Konig HH, Bienert F, Brinkmann J, Herbarth L, Kramer E, Steinisch P, Freudenstein F, Terhalle R, Grosse Y, Bock S, Posselt J, Beutel C, Reif F, Kirchhoff F, Neuschwander C, Loffler F, Brunner L, Dickmeis P, Heidenthal T, Schmitz L, Chase DP, Seelenmeyer C, Alscher MD, Tegtbur U, Dirmaier J. Telephone health coaching with exercise monitoring using wearable activity trackers (TeGeCoach) for improving walking impairment in peripheral artery disease: study protocol for a randomised controlled trial and economic evaluation. BMJ Open. 2020 Jun 4;10(6):e032146. doi: 10.1136/bmjopen-2019-032146. PMID 32503866

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT03496948/Prot_SAP_002.pdf